CLINICAL TRIAL: NCT02698995
Title: Analgetic Efficiency of Single-shot Perineural Low Dose Dexamethasone Added to Infraclavicular Block Anesthesia for Upper Limb Surgery
Brief Title: Perineural Low-dose Dexamethasone Added to Infraclavicular Block Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foisor Orthopedics Clinical Hospital (Other)
Responsible Party: Principal Investigator, Munteanu Ana Maria, MD, PhD, MD PhD, Foisor Orthopedics Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID AN-002-14
Record Dates: First submitted 2016-02-19; First posted 2016-03-04 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Calcium Dobesilate; Ropivacaine; Acetaminophen; Morphine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Placebo Comparator): VIB block with ropivacaine 0,5%100 mg+lidocaine1%100 mg+1 ml saline=21 ml. After the block regression, at the first analgetic request the patients received the analgesia protocol was started for 24 h with paracetamol 1 g IV every 8 h and lornoxicam 8 mg PO every 12 h; if VAS was still over 3 after 30 min, morphine was given as a loading bolus of 0.05 mg/kg IV supplemented with 2 mg IV every 5 minutes until VAS <3. After 2 h morphine was administered SC ½ of the total loading dose at request.
  Interventions: Drug: Ropivacaine; Drug: Paracetamol; Drug: Morphine; Drug: Lidocaine
- Group B (Active Comparator): VIB block with ropivacaine 0,5%100 mg+lidocaine1%100 mg+2 mg dexamethasone=21 ml. After the block regression, at the first analgetic request the patients received the analgesia protocol was started for 24 h with paracetamol 1 g IV every 8 h and lornoxicam 8 mg PO every 12 h; if VAS was still over 3 after 30 min, morphine was given as a loading bolus of 0.05 mg/kg IV supplemented with 2 mg IV every 5 minutes until VAS <3. After 2 h morphine was administered SC ½ of the total loading dose at request.
  Interventions: Drug: Dexamethasone; Drug: Ropivacaine; Drug: Paracetamol; Drug: Morphine; Drug: Lidocaine
- Group C (Active Comparator): VIB block with ropivacaine 0,5%100 mg+lidocaine1%100 mg+4 mg dexamethasone=21 ml. After the block regression, at the first analgetic request the patients received the analgesia protocol was started for 24 h with paracetamol 1 g IV every 8 h and lornoxicam 8 mg PO every 12 h; if VAS was still over 3 after 30 min, morphine was given as a loading bolus of 0.05 mg/kg IV supplemented with 2 mg IV every 5 minutes until VAS <3. After 2 h morphine was administered SC ½ of the total loading dose at request.
  Interventions: Drug: Dexamethasone; Drug: Ropivacaine; Drug: Paracetamol; Drug: Morphine; Drug: Lidocaine

INTERVENTIONS:
Drug: Dexamethasone — One hour before surgery the patients received single shot VIB block with the mixture according to the group allocation
  Other Names: Decadron
  Arms: Group B; Group C
Drug: Ropivacaine — One hour before surgery the patients received single shot VIB block with the mixture according to the group allocation
  Other Names: Naropin
Drug: Paracetamol — After the block regression, at the first analgetic request the patients received the same analgesia protocol
  Other Names: Perfalgan
Drug: Morphine — After the block regression, at the first analgetic request the patients received the same analgesia protocol
  Other Names: Morphine Sulfate ER
Drug: Lidocaine — One hour before surgery the patients received single shot VIB block with the mixture according to the group allocation
  Other Names: Xylocaine

SUMMARY:
Dexamethasone has an evidence-based indication in postoperative emesis prophylaxy and as a antiinflammatory steroid. Although the perineural administration is off-label, several studies recognised its analgetic action as an adjuvant for peripheral nerves blockade, permitting to reduce the concentration of the local anesthetics and extending the sensory and motor block.Questions remain concerning the mechanism of action, optimal dose, the lack/degree of toxicity and the comparison with intravenous administration.The aim of this prospective randomized controlled study is to investigate the efficacy of analgesia with 4 mg or 2 mg Dexamethasone added to a combination of ropivacaine 0,5% and lidocaine 1% in vertical infraclavicular blockade (VIB) anesthesia for upper limb surgery.

DETAILED DESCRIPTION:
The investigators conducted a prospective randomized controlled study in 150 patients American Society of Anesthesiologists (ASA) score I-III scheduled for upper limb surgery , divided in 3 groups: group A received anesthesia VIB block with ropivacaine 0,5% 100 mg +lidocaine 1%+1 ml saline; group B received VIB block with ropivacaine 0,5% 100 mg +lidocaine 1% + 2 mg dexamethasone; group C received ropivacaine 0,5% 100 mg +lidocaine 1% + 4 mg dexamethasone.The anesthesiologist may use the ultrasound for visual guidance, but should also use the nerve stimulator in order to maintain the homogeneity of the procedure.

Intraoperative sedation was provided with intermittent bolus 10-20 mg IV Propofol. Postoperatively all patients received the same analgetic protocol when Visual Analog Pain Scale (VAS) over 3 with IV Perfalgan and Lornoxicam 8 mg/12 hours for 24 hours. If after 30 minutes VAS is still over 3, a loading dose of morphine 0,05 mg/kg should be administered. At first analgetic request, the nurse conducts an ice-probe test to both arms and will note the answer: same cold, slightly burn, burn, aching with the reason to test the potentially hyperalgesia effect related to ropivacaine. The data recorded are: time to first analgetic use, VAS at block regression, ice-probe test, motor and sensitive block duration, glycemic variations at 4 h, neurological complications immediately after block, total morphine consumption.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III,
* BMI<40,
* non-anemic

Exclusion Criteria:

* High risk grade hypertension, chronic renal failure, known allergy to local anesthetic or NSAIDs, chronic treatment with steroids, drugs dependency, history of diabetes mellitus, ulcer or chronic gastritis, infection on the puncture site, chronic obstructive pulmonary disease, neuropathy at the surgical level

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Sensory block duration | First 24 hours
  The time in minutes measured between VIB block to first analgetic request

SECONDARY OUTCOMES:
Motor block duration | First 24 hours postoperatively
  The time in minutes measured between VIB block to complete movement of the hand
Glycemic variations at 4 hours post-VIB block | First 4 hours postoperatively
  Determination of blood sugar level
Number of patients opioid free analgesia | First 24 hours postoperatively
  Number of reported patients with no need opioid analgesia
VAS at the block regression | First 24 hours postoperatively
  VAS evaluation on the VAS scale (0 - no pain, 10 - the worst pain possible )
Cutaneous temperature ice-probe | First 24 hours postoperatively
  The cold sensation on ice-probe test to both arms could be the same or burn likely
Total morphine consumption at 24 hours | First 24 hours postoperatively
  Cumulative morphine administration in milligrams

CONTACTS AND LOCATIONS:
Overall Officials: Ioan Cristian Stoica, MD Prof, Study Director — Foisor Orthopedics Clinical Hospital
Locations (1):
- Foisor Orthopedic Clinical Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kalichman MW, Powell HC, Myers RR. Pathology of local anesthetic-induced nerve injury. Acta Neuropathol. 1988;75(6):583-9. doi: 10.1007/BF00686203. PMID 3376761
- [Result] Myers RR, Kalichman MW, Reisner LS, Powell HC. Neurotoxicity of local anesthetics: altered perineurial permeability, edema, and nerve fiber injury. Anesthesiology. 1986 Jan;64(1):29-35. PMID 3942334
- [Result] Zink W, Graf BM. The toxicity of local anesthetics: the place of ropivacaine and levobupivacaine. Curr Opin Anaesthesiol. 2008 Oct;21(5):645-50. doi: 10.1097/ACO.0b013e32830c214c. PMID 18784493
- [Result] Williams BA, Hough KA, Tsui BY, Ibinson JW, Gold MS, Gebhart GF. Neurotoxicity of adjuvants used in perineural anesthesia and analgesia in comparison with ropivacaine. Reg Anesth Pain Med. 2011 May-Jun;36(3):225-30. doi: 10.1097/AAP.0b013e3182176f70. PMID 21519308
- [Result] Huynh TM, Marret E, Bonnet F. Combination of dexamethasone and local anaesthetic solution in peripheral nerve blocks: A meta-analysis of randomised controlled trials. Eur J Anaesthesiol. 2015 Nov;32(11):751-8. doi: 10.1097/EJA.0000000000000248. PMID 25774458
- [Result] Kawanishi R, Yamamoto K, Tobetto Y, Nomura K, Kato M, Go R, Tsutsumi YM, Tanaka K, Takeda Y. Perineural but not systemic low-dose dexamethasone prolongs the duration of interscalene block with ropivacaine: a prospective randomized trial. Local Reg Anesth. 2014 Apr 5;7:5-9. doi: 10.2147/LRA.S59158. eCollection 2014. PMID 24817819